CLINICAL TRIAL: NCT00805675
Title: A Randomized, Open-label, Controlled, Exploratory Trial to Characterize the Results of Daily Oral Administration of Telbivudine 600 mg and Tenofovir Disproxil Fumarate 300 mg in Combination or Telbivudine 600 mg or Tenofovir Disproxil Fumarate 300 mg Monotherapy Given Over 12 Weeks on the Kinetics of Hepatitis B Virus DNA in Adults With HBeAg Positive Compensated CHB
Brief Title: Effects of Telbivudine and Tenofovir Disoproxil Fumarate Treatment on the Hepatitis B Virus DNA Kinetics in CHB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AHK01
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-01

CONDITIONS: Hepatitis B Virus
Keywords: Chronic HBV; Asian adult subjects with chronic HBV, in immune tolerant phase, and positive for hepatitis B e antigen (HBeAg)
MeSH Terms: conditions — Hepatitis B | interventions — Telbivudine; Tenofovir

ARMS (3):
- Telbivudine 600 mg monotherapy (Experimental): All patients in this arm were randomized to receive Telbivudine (LDT) 600 mg QD. Patients were randomized prior to the first dose of study medication, which was defined as the study Baseline (Day 1) Visit. Subsequently, patients returned to the clinic at Days 2, 4, 6, 8, 11, 15 (Wk 2), 22 (Wk 3), 29 (Wk 4), 43 (Wk 6), 57 (Wk 8), and 85 (Wk 12) during the 12 weeks treatment phase.
  Interventions: Drug: Telbivudine
- Tenofovir disproxil fumarate 300 mg monotherapy (Active Comparator): All patients in this arm were randomized to receive Tenofovir disoproxil fumarate 300 mg(equivalent to tenofovir disoproxil 245 mg)QD. Patients were randomized prior to the first dose of study medication, which was defined as the study Baseline (Day 1) Visit. Subsequently, patients returned to the clinic at Days 2, 4, 6, 8, 11, 15 (Wk 2), 22 (Wk 3), 29 (Wk 4), 43 (Wk 6), 57 (Wk 8), and 85 (Wk 12) during the 12 weeks treatment phase.
  Interventions: Drug: Tenofovir
- Telbivudine 600 mg and Tenofovir 300 mg (Active Comparator): All patients in this arm were randomized to receive Telbivudine (LDT) 600 mg QD and Tenofovir (TDF) 300 mg (equivalent to Tenofovir disoproxil 245 mg)QD. Patients were randomized prior to the first dose of study medication, which was defined as the study Baseline (Day 1) Visit. Subsequently, patients returned to the clinic at Days 2, 4, 6, 8, 11, 15 (Wk 2), 22 (Wk 3), 29 (Wk 4), 43 (Wk 6), 57 (Wk 8), and 85 (Wk 12) during the 12 weeks treatment phase.
  Interventions: Drug: Telbivudine plus tenofovir

INTERVENTIONS:
Drug: Telbivudine — 600 mg monotherapy supplied in film-coated tablets.
  Arms: Telbivudine 600 mg monotherapy
Drug: Tenofovir — Tenofovir disoproxil fumarate was supplied in 300 mg tablets
  Arms: Tenofovir disproxil fumarate 300 mg monotherapy
Drug: Telbivudine plus tenofovir — Telbivudine 600 mg and Tenofovir 300 mg were purchased in commercial packs. Patients were instructed to take medication(s) orally every morning either with or without food.
  Arms: Telbivudine 600 mg and Tenofovir 300 mg

SUMMARY:
The purpose of this study is to compare the safety, tolerability and effectiveness of 12 weeks of treatment with telbivudine 600 mg daily plus tenofovir DF 300 mg one daily (OD) taken together vs. tenofovir DF 300 mg once daily (QD) or vs telbivudine 600 mg monotherapy daily (QD). This is an open labeled, active controlled, viral kinetics study which means the subjects and study doctor will know what study drug subjects have been assigned. This study is open to male and female subjects, <40 years of age, who have been infected with HBV for at least 6 months and have not received oral treatment for HBV.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection, defined as positive serum HBsAg for at least 6 months, or HBsAg positive > 3 months and negative for IgM anti-HBc and positive for IgG anti-HBc
* Age < 40 years old
* HBeAg positive
* HBV DNA > or = to 10^7 copies/mL by Abbott real-time PCR
* ALT < or = to 1 ULN
* Willing and able to provide written informed consent
* No prior oral HBV therapy (e.g., nucleotide and/or nucleoside therapy or other investigational agents for HBV infection)
* Is willing and able to comply with the study drug regimen and all other study procedures and requirements
* Is willing and able to provide written informed consent before any study assessment is perform

Exclusion Criteria:

* Decompensated liver disease defined as direct (conjugated) bilirubin > 1.2 × ULN, PT > 1.2 × ULN, platelets < 150,000/mm3, serum albumin < 3.5 g/dL, or prior history of clinical hepatic decompensation (e.g. ascites, jaundice, encephalopathy, variceal hemorrhage).
* Received interferon (pegylated or not) therapy within 6 months of the screening visit
* α-fetoprotein > 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* Co-infection with HCV (by serology), or HIV,
* Significant renal, cardiovascular, pulmonary, or neurological disease.
* Received solid organ or bone marrow transplantation.
* Is currently receiving therapy with immunomodulators (e.g., corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion.
* Has proximal tubulopathy.
* Use of other investigational drugs at the time of enrollment, or within 30 days
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Is pregnant or breastfeeding.
* Is a women of child-bearing potential (WOCBP)unless post-menopausal or using one or more acceptable method of contraception.
* Patient has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study.
* Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years.
* Patient has a medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Department of Medicine, Queen Mary Hospital, Hong Kong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 participants signed informed consent. 36 patients were not recruited. 32 patients failed inclusion/exclusion criteria and 4 withdrew consent. 47 participants were eligible and recruited.
Pre-assignment Details: Out of a total enrollment of 47 participants, 1 participant withdrew consent before being randomized into treatment.
Groups:
- Telbivudine 600 mg Monotherapy: All patients in this arm were randomized to receive Telbivudine (LDT) 600 mg QD. Patients were randomized prior to the first dose of study medication, which was defined as the study Baseline (Day 1) Visit. Subsequently, patients returned to the clinic at Days 2, 4, 6, 8, 11, 15 (Wk 2), 22 (Wk 3), 29 (Wk 4), 43 (Wk 6), 57 (Wk 8), and 85 (Wk 12) during the 12 weeks treatment phase. Furthermore, patients scheduled to Post-treatment Follow-up visits at Day 113 (Wk 16), Day 141 (Wk 20), and Day 169 (Wk 24) . At each of these visits routine tests and adverse event inquiry were performed.
- Tenofovir Disproxil Fumarate 300 mg Monotherapy: All patients in this arm were randomized to receive Tenofovir disoproxil fumarate 300 mg(equivalent to tenofovir disoproxil 245 mg)QD. Patients were randomized prior to the first dose of study medication, which was defined as the study Baseline (Day 1) Visit. Subsequently, patients returned to the clinic at Days 2, 4, 6, 8, 11, 15 (Wk 2), 22 (Wk 3), 29 (Wk 4), 43 (Wk 6), 57 (Wk 8), and 85 (Wk 12) during the 12 weeks treatment phase. Furthermore, patients scheduled to Post-treatment Follow-up visits at Day 113 (Wk 16), Day 141 (Wk 20), and Day 169 (Wk 24) . At each of these visits routine tests and adverse event inquiry were performed.
- Telbivudine 600 mg and Tenofovir 300 mg: All patients in this arm were randomized to receive Telbivudine (LDT) 600 mg QD and Tenofovir (TDF) 300 mg (equivalent to Tenofovir disoproxil 245 mg)QD. Patients were randomized prior to the first dose of study medication, which was defined as the study Baseline (Day 1) Visit. Subsequently, patients returned to the clinic at Days 2, 4, 6, 8, 11, 15 (Wk 2), 22 (Wk 3), 29 (Wk 4), 43 (Wk 6), 57 (Wk 8), and 85 (Wk 12) during the 12 weeks treatment phase. Furthermore, patients scheduled to Post-treatment Follow-up visits at Day 113 (Wk 16), Day 141 (Wk 20), and Day 169 (Wk 24) . At each of these visits routine tests and adverse event inquiry were performed.
Period: Overall Study
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Started | 16 | 14 | 16
Completed | 16 | 14 | 15
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg | Total
Number analyzed (Participants) | 16 | 14 | 16 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.58) | 27.3 (4.94) | 28.9 (5.55) | 28.1 (6.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 10 | 22
  Male | 9 | 9 | 6 | 24
Region of Enrollment [Number; unit: participants]
  China | 16 | 14 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Level From Baseline to Week 12.
Description: Baseline HBV DNA is defined as the last pre-dose assessment of HBV DNA. Serum HBV DNA determinations were performed at a central laboratory through use of the COBAS TaqMan™ HBV DNA assay (Roche Molecular Systems, Pleasanton, CA, USA) which utilized the Real-time polymerase chain reaction (PCR) method and automated extraction by Cobas Ampliprep (threshold for detection 12 IU/mL). The Screening serum HBV DNA values must be ≥ 7 log10 copies/mL by COBAS TaqMan™ HBV DNA assay.
Time Frame: Baseline, Week 12
Population: The Intent to Treat (ITT) data set consisted of the participants that had been randomized and had taken the investigational drug at least once.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
log10 copies/mL | -3.852 (0.9330) | -4.175 (0.7476) | -4.374 (0.9774)

2. Secondary Outcome: Change in Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Level From Baseline to Weeks 2, 4 and 8.
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
log10 copies/mL
  Week 2 | -2.657 (0.6683) | -2.541 (0.4876) | -2.689 (0.5951)
  Week 4 | -2.985 (0.8019) | -3.060 (0.6230) | -3.225 (0.8149)
  Week 8 | -3.474 (0.8829) | -3.621 (0.6737) | -3.845 (0.849)

3. Secondary Outcome: Percentage of Patients Who Are Polymerase Chain Reaction(PCR)Negative at Week 12
Description: Polymerase Chain Reaction (PCR) Negative is defined as HBV DNA levels <25 copies/ml.
Time Frame: Week 12
Population: The Intent to Treat (ITT) data set consisted of the participants that had been randomized and had taken the investigational drug at least once. (1 pat DNA<169 cps/ml)
Measure: Number; unit: Percentage of Participants
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Percentage of Patients Who Achieve Hepatitis B "e" Antigen (HBeAg) Loss and HBeAg Seroconversion at Week 12
Description: HBeAg loss is defined as the loss of detectable serum HBeAg in a patient who was HBeAg positive at baseline. HBeAg seroconversion is defined as HBeAg loss with detectable Hepatitis B 'e' antibody (HBeAb). HBeAg stands for hepatitis B "e" antigen. This antigen is a protein from the hepatitis B virus that circulates in infected blood when the virus is actively replicating. The presence of HBeAg suggests that the person is infectious and is able to spread the virus to other people.
Time Frame: Week 12
Population: The Intent to Treat (ITT) data set consisted of the participants that had been randomized and had taken the investigational drug at least once. Note: In this analysis 1 patient HBeAg loss in the Telbivudine 600 mg and Tenofovir 300 mg Treatment Group.
Measure: Number; unit: Percentage of Participants
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
Percentage of Participants | 0 | 0 | 0

5. Secondary Outcome: Characterization of Very Early Viral Kinetics Through Estimated Viral Load
Description: The underlying bi-phasic model of viral kinetics can be described as follows:
  V(t) (1 )pI(t) cV(t)I(t) (1 ) (T I(t))V(t) I(t)where V denotes serum viral load, I productively infected cells, ε the efficiency factor of blocking virus production, p the viral production rate, c the viral clearance rate, η the efficiency factor of blocking de novo infection, β the de novo infection rate, Tg comprise all infected and uninfected target cells, and δ the rate of infected cell loss
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
log10 copies/ml | 8.9 (0.6) | 8.7 (0.8) | 8.7 (0.6)

6. Secondary Outcome: Characterization of Very Early Viral Kinetics Through Viral Clearance
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day^-1
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
day^-1 | 0.98 (0.19) | 1.19 (0.62) | 1.08 (0.75)

7. Secondary Outcome: Characterization of Very Early Viral Kinetics Through Rate of Infected Cell Loss
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day^-1
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
day^-1 | 0.04 (0.01) | 0.06 (0.02) | 0.05 (0.02)

8. Secondary Outcome: Characterization of Very Early Viral Kinetics Through Efficiency Factor of Blocking Virus Production.
Description: The underlying bi-phasic model of viral kinetics can be described as follows:
  V(t) (1 )pI(t) cV(t) I(t) (1 ) (T I(t))V(t) I(t) where V denotes serum viral load, I productively infected cells, ε the efficiency factor of blocking virus production, p the viral production rate, c the viral clearance rate, η the efficiency factor of blocking de novo infection, β the de novo infection rate, Tg comprise allinfected and uninfected target cells, and δ the rate of infected cell loss
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
Percentage | 98.8 (1.9) | 99.0 (1.3) | 99.1 (0.8)

9. Secondary Outcome: Characterization of Very Early Viral Kinetics Through Half-live of Free Virus
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Number analyzed (Participants) | 16 | 14 | 16
Hours | 18.1 (4.4) | 16.4 (5.8) | 18.9 (6.9)

ADVERSE EVENTS:
Arm/Group | Telbivudine 600 mg Monotherapy | Tenofovir Disproxil Fumarate 300 mg Monotherapy | Telbivudine 600 mg and Tenofovir 300 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 8/14 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telbivudine 600 mg Monotherapy (N=16) | Tenofovir Disproxil Fumarate 300 mg Monotherapy (N=14) | Telbivudine 600 mg and Tenofovir 300 mg (N=16)
Dizziness (Cardiac disorders) | 0 | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Influenza like illness (General disorders) | 4 | 2 | 0
Exercise tolerance descreased (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 5 | 3 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.